CLINICAL TRIAL: NCT04475458
Title: Pediatric Ultrasound-guided Dorsal Penile Nerve Block Plus Sedation in Spontaneous Breathing: An Observational Study
Brief Title: Pediatric Ultrasound-guided Dorsal Penile Nerve Block Plus Sedation in Spontaneous Breathing
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Luigi Vetrugno, Prof., Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: Ultrasound guided DPNB
Record Dates: First submitted 2020-07-10; First posted 2020-07-17 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Child, Only
Keywords: dorsal nerve penis block; sedation; spontaneous breathing; circumcision; pediatric surgery; ultrasound guided

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LANDMARK: The children who underwent circumcision received general anesthesia plus dorsal penis nerve block performed by the surgeon with a landmark technique.
- ULTRASOUND: The children who underwent circumcision received sedation (in spontaneous breathing) plus ultrasound-guided dorsal penis nerve block.
  Interventions: Procedure: Ultrasound-guided dorsal penile nerve block

INTERVENTIONS:
Procedure: Ultrasound-guided dorsal penile nerve block — This block is performed by the anesthesiologist, after sedation. With an in-plane approach, the tissues around the dorsal penis nerves are visualized. The needle has to pass through Buck's fascia and there the local anesthetic is released.
  Groups: ULTRASOUND

SUMMARY:
One of the most frequent surgical procedures in the pediatric population is circumcision, following which postoperative pain could be stressful. Usually, the most common approach is combining regional anesthesia techniques such as landmark dorsal penile nerve block (DPNB) with general anesthesia (GA). The hypothesis of this study investigates ultrasound-guided DPNB plus sedation in spontaneous breathing.

ELIGIBILITY:
Inclusion Criteria:

* candidates to circumcision
* age between 6 months and 17 years
* American Society of Anesthesiologists (ASA) physical status < 3
* written consent of the parents

Exclusion Criteria:

* allergies to local anesthetics
* younger than 6 months and older than 17 years
* ASA physical status =/> 3
* no written consent of the parents

Ages: 6 Months to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients' anthropometric data were collected. Data related to the anesthetic technique, pharmacological therapy, vital parameters were registered as well as the time to discharge from the operatory room to the post-anesthesia care unit.
  Opioid consumption and nonsteroidal anti-inflammatory drugs during and after surgery were noted. Pain and complications immediately after surgery, at 4 and 72 hours after surgery were registered.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Time to discharge | 1 hour after end of surgery
  The time to discharge from the operating room to the post-anesthesia care unit is measured and compared between the two groups.

SECONDARY OUTCOMES:
Number of patients needed ventilation | 1 hour after beginning of surgery
  Patients who received general anesthesia where all ventilated mechanically. In the ultrasound group, patients maintained spontaneous breathing and were noted the ones who needed ventilation.
Opioid sparing | 1 hour after beginning of surgery
  The dosage of opioids were measured and compared between the two groups.
Postoperative pain | Immediately after surgery, 4 and 72 hours after surgery
  Pain levels were compared between the two groups with the Faces, Legs, Activity, Cry and Consolability (FLACC) scale for children < 3 years (a score between 0 and 3 corresponds to a slight pain, in the range 4-7 to moderate pain and score> 7 to a severe pain), faces pain scale for children between 3 e 8 years (the scale shows a series of faces ranging from a happy face or no hurt at score 0, to a crying face at score 10, which represents "hurts like the worst pain imaginable", the patient chooses the face that best describes their level of pain) and the numerical rate scale (NRS) for children > 8 years-old (patients are asked to circle the number between 0 and 10 that fits best to their pain intensity, zero represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'). Analgesics and nonsteroidal anti-inflammatory drugs were registered in the two groups.
Complications | Immediately after surgery, 4 and 72 hours after surgery
  Postoperative complications were analyzed and compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Intensive Care Clinic - Department of Medicine - ASUIUD, Udine, Italy

REFERENCES:
- [Background] Cyna AM, Middleton P. Caudal epidural block versus other methods of postoperative pain relief for circumcision in boys. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD003005. doi: 10.1002/14651858.CD003005.pub2. PMID 18843636
- [Background] Suleman MI, Akbar Ali AN, Kanarek V, Li M, Patel A. Ultrasound Guided In-Plane Penile Nerve Block for Circumcision: A New, Modified Technique Suggests Lower Anesthetic Volume and Narcotic Use. Middle East J Anaesthesiol. 2016 Oct;23(6):647-53. PMID 29939703
- [Background] Sandeman DJ, Dilley AV. Ultrasound guided dorsal penile nerve block in children. Anaesth Intensive Care. 2007 Apr;35(2):266-9. doi: 10.1177/0310057X0703500217. PMID 17444318
- [Background] O'Sullivan MJ, Mislovic B, Alexander E. Dorsal penile nerve block for male pediatric circumcision--randomized comparison of ultrasound-guided vs anatomical landmark technique. Paediatr Anaesth. 2011 Dec;21(12):1214-8. doi: 10.1111/j.1460-9592.2011.03722.x. PMID 22023417
- [Derived] Dottore B, Meroi F, Tomasino S, Orso D, Comuzzi M, Vernaccini N, Vetrugno L, Intini S, Bove T. Pediatric ultrasound-guided dorsal penile nerve block and sedation in spontaneous breathing: a prospective observational study. Front Med (Lausanne). 2023 Dec 4;10:1268594. doi: 10.3389/fmed.2023.1268594. eCollection 2023. PMID 38116040